CLINICAL TRIAL: NCT06639945
Title: Clinical Trail of Transcranial MR-guided Focused Ultrasound in the Treatment of Motor Symptoms in Patients with Parkinson' Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhengguo Liu, Department of Neurology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XHEC-C-2024-125-2-1
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease, Idiopathic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum stimulation followed by Sham stimulation (Experimental)
  Interventions: Device: transcranial MR-guided focused ultrasound
- Sham stimulation followed by Verum stimulation (Experimental)
  Interventions: Device: transcranial MR-guided focused ultrasound

INTERVENTIONS:
Device: transcranial MR-guided focused ultrasound — MRI-guided transcranial focused ultrasound (MRgFUS) combines magnetic resonance imaging (MRI) with focused ultrasound to target specific areas in the brain non-invasively. MRgFUS allows for treatment without surgical incisions, leading to fewer risks and a quicker recovery. MRI provides real-time imaging that helps precisely locate and treat affected brain regions, such as the thalamus or globus pallidus.The procedure allows for continuous monitoring of the treatment effects, enabling adjustments as needed.

SUMMARY:
Randomized, double-blind, self-cross-over control (After the first visit, patients are divided into two groups, randomly receiving real stimulation/placebo stimulation. 10 days later, during the second visit, a cross-over occurs: patients who received real stimulation in the first visit will receive placebo stimulation in the second visit, and vice versa. The grouping situation remains blinded for the patients, TMS analysts, and video analysts.)

ELIGIBILITY:
Inclusion Criteria:

* Meets the clinical probable Parkinson's disease diagnostic criteria proposed by MDS-UPDRS;
* Disease duration of 4 years or less;
* Unmedicated or has been off medication for more than 12 hours, with H&Y stage ≤ 2.

Exclusion Criteria:

* History of stroke or seizures, dementia; previous surgical interventions for Parkinson's disease; contraindications for TMS (such as cardiac pacemakers, transcranial implants, and metal implants); severe mental disorders such as depression or psychosis; inability to understand the study procedures; use of antipsychotic medications; pregnancy.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
UPDRS-III | 2 weeks and 4 weeks
  Change in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score of part III from Day 1 to 1 year. The part III of the MDS-UPDRS assess motor function in best on phase. The score range is 0-132, where a higher score means more severe motor impairment.

SECONDARY OUTCOMES:
TMS parameters | 2 weeks and 4 weeks
  Resting Motor Threshold, Input-Output Curve, Cortical Silent Period, Short-latency Afferent Inhibition, SAI, Interhemispheric Inhibition, Long-term Potentiation.
cortical activation detected by fNIRS | 2 weeks and 4 weeks
  Using near-infrared brain imaging systems, have patients perform finger tapping, fist clenching, and forearm rotation movements to observe brain region activation.